CLINICAL TRIAL: NCT06032117
Title: Characterizing Protein Biomarkers of Post-infection Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Other Study IDs: 1891300
Record Dates: First submitted 2023-07-28; First posted 2023-09-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Post-infectious Irritable Bowel Syndrome; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Approximately 6 ml of blood will be collected from each participant. Samples will be centrifuged (1,000-2,000 x g for 10 minutes), the serum separated and placed into an Eppendorf tube/cryovials, and stored in a -80 °C fridge until analysis. The proteomics lab will use 100ul of serum, and the rest will be banked in cryovials. The de-identified samples will be stored in a fridge at UNR, which is in a locked room and accessible only to the University of Nevada, Reno (UNR) research team. The researchers will not identify these samples or perform identifying tests (e.g., genetics tests) on those samples. The samples will be stored for a period of 3 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post infectious irritable bowel syndrome group: Participants will have post-infectious IBS (as identified via Rome IV criteria or previous physician diagnosis)
- Healthy control group: Participants will not have post-infectious IBS, matched on age group, sex, and race/ethnicity.
- Irritable bowel syndrome group: Participants will have IBS, matched on age group, sex, and race/ethnicity.

SUMMARY:
The investigators will characterize and compare protein signatures between groups with and without post-infection irritable bowel syndrome (PI-IBS). From previous Healthy Nevada Project (HNP) participants, at least 60 patients with PI-IBS and 60 healthy controls will undergo additional proteomics testing, age, sex and race/ethnicity-matched healthy. The investigators will use proteomic testing to detect, quantify and characterize serum protein biomarkers and protein signatures, and compare biomarkers and signatures between the patient groups of interest. Serum samples will be analyzed by the Nevada Proteomics Center. Samples will first undergo protein digestion, then peptides are separated using liquid chromatography (LC), mass spectral analysis is performed using an Orbitrap Eclipse mass spectrometer (Thermo Scientific, San Jose, CA) using data-independent acquisition (DIA). Library generation and data analysis will be performed using Spectronaut software (Biognosys, Schlieren, Switzerland). The Nevada Proteomics Center and Bioinformatics Center will be engaged during the data analyses comparing biomarkers and signatures between the patient groups of interest. This research aim has the potential to add to our understanding of the underlying mechanisms of PI-IBS and to create reliable differentiating protein biomarkers to better diagnose PI-IBS.

DETAILED DESCRIPTION:
The investigators will characterize and compare protein signatures between groups with and without PI-IBS. From previous HNP participants, at least 60 patients with PI-IBS and 60 healthy controls will be recruited to undergo additional proteomics testing, age, sex and race/ethnicity-matched healthy. The investigators will use proteomic testing to detect, quantify and characterize serum protein biomarkers and protein signatures, and compare biomarkers and signatures between the patient groups of interest. Serum samples will be analyzed by the Nevada Proteomics Center. Samples will first undergo protein digestion, then peptides are separated using liquid chromatography (LC), mass spectral analysis is performed using an Orbitrap Eclipse mass spectrometer (Thermo Scientific, San Jose, CA) using data-independent acquisition (DIA). Library generation and data analysis will be performed using Spectronaut software (Biognosys, Schlieren, Switzerland). The Nevada Proteomics Center and Bioinformatics Center will be engaged during the data analyses comparing biomarkers and signatures between the patient groups of interest. This research aim has the potential to add to our understanding of the underlying mechanisms of PI-IBS and to create reliable differentiating protein biomarkers to better diagnose PI-IBS.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a Healthy Nevada Project record and linked Renown Health medical record
* Must be between 18 and 89 years of age
* Must have previously consented to being contacted and have updated contact information

Exclusion Criteria:

-None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To approximate the population of Washoe county in our recruitment survey we will use a stratified random sampling scheme to randomly sample from strata of sex and ethnicity from within the HNP, so that our study sample is approximately 50% male and 50% female, and approximately 24.5% Hispanic. From these survey responses, the PI will be able to find 60 PI-IBS cases, and 60 controls. We will send the recruitment email to additional participants following the same methods described above (e.g., batching 1000 potential participants at a time, oversampling Hispanics and women in the same way) until we have found 60 total PI-IBS participants. If we have further difficulties finding PI-IBS participants, we may send targeted emails to previous HNP participants who has an ICD 10 code indicating a gastrointestinal infection or IBS in the last 5 years.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Rome IV diagnosis of post-infectious irritable bowel syndrome | Day 1
  Rome IV is used to diagnose IBS, and participants must additionally have had sudden onset of their IBS with either 1) IBS symptoms developing immediately AFTER foreign travel/deployment or 2) immediately AFTER acute infectious gastroenteritis with two or more of: fever, vomiting, diarrhea

SECONDARY OUTCOMES:
Participant-reported post-infectious irritable bowel syndrome | Day 1
  Participants report that they have been diagnosed with IBS by a physician and that they still have symptoms, and participants must additionally have had sudden onset of their IBS with either 1) IBS symptoms developing immediately AFTER foreign travel/deployment or 2) immediately AFTER acute infectious gastroenteritis with two or more of: fever, vomiting, diarrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Renow Health, Mae Anne Clinic, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Final study results will be posted to ClinicalTrials.gov within 12 months of study completion.
  The study protocol and statistical analysis plans will be shared on Open Science Framework (OSF) before the first biological samples are collected.
  The informed consent form will be posted to OSF within 60 days of the last study visit by any participant.
  Analytic code and relevant data will be posted to OSF upon publication of study results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
URL: https://osf.io/2z4rj/